CLINICAL TRIAL: NCT00663494
Title: MMP is Produced in Failing Hearts
Brief Title: Matrix Metalloproteinase (MMP) in Heart Failure
Status: Completed | Type: Observational
Sponsor: Tottori University Hospital (Other)
Responsible Party: Kazuhide Ogino, Tottori University Hospital
Other Study IDs: #244
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2008-04

CONDITIONS: Chronic Stable Heart Failure
Keywords: heart failure; MMP; coronary sinus
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the production of MMP in failing hearts.

DETAILED DESCRIPTION:
Myocardial fibrosis is observed in failing hearts and parallel to the progression of chronic heart failure (CHF) and myocardial remodeling. Matrix metalloproteinases (MMPs) are considered markers of fibrosis. Recently, circulating MMPs can be measured and are elevated in patients with CHF. However, MMPs it is still unclear whether MMPs are produced in failing hearts. Thus, the purpose of this study is to evaluate the production of MMP in failing hearts.

ELIGIBILITY:
Inclusion Criteria:

* chronic stable heart failure

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: chronic heart failure
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2003-02; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
MMPs level of coronary sinus